CLINICAL TRIAL: NCT05413070
Title: Improving Performance on Choosing Wisely Low Back Pain Measures in Primary Care: Learning From Within
Brief Title: Quality Improvement re: Choosing Wisely Back Pain Measures
Acronym: SCV LBP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Center for Health Innovation (Unknown)
Responsible Party: Principal Investigator, Michelle Rockwell, Senior Research Associate, Carilion Clinic
Other Study IDs: IRB-22-1568
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Back Pain, Low; Back Pain; Back Pain Lower Back Chronic
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Low-Value Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lowest Performing Practices: This is the group of 5 to 10 primary care practices that incurred the highest amount of low-value back pain imaging based on claims data reports. This group will receive the survey and the intervention (brief training sessions in existing quality improvement meetings, performance reports, etc.).
  Interventions: Behavioral: Multimodal approach to QI for Low-Value Care
- Highest Performing Practices: This is the group of 5 primary care practices that incurred the lowest amount of low-value back pain imaging based on claims data reports. This group will only receive the survey.

INTERVENTIONS:
Behavioral: Multimodal approach to QI for Low-Value Care — Up to 4 brief educational components in existing quality meetings Informational email/newsletter Individualized performance feedback reports Educational resources for patients
  Groups: Lowest Performing Practices

SUMMARY:
As

DETAILED DESCRIPTION:
Two common low-value services are related to acute low back pain. Choosing Wisely advises avoiding the use of imaging during the first 6 weeks of low back pain (per the American Academy of Family Physicians and other organizations). Similarly, Choosing Wisely advises avoiding opioids in the treatment of low back pain until other alternatives have been attempted (per the North American Spine Society). Together, overutilization of these two services (imaging and opioids for low back pain) costs more than $500 annually, not including downstream costs, and is a source of patient harm. In the state of Virginia, the Virginia Center for Health Innovation has identified the two back pain measures as priority for reducing as part of their 3-year intervention (Smarter Care Virginia): https://www.vahealthinnovation.org/scv/

As a participant in Smarter Care Virginia (SCV), Carilion receives data showing each Carilion Clinic clinician's performance on SCV measures, including the two back pain measures. For example, Carilion receives a database that lists the clinician's name, department, number of appropriate orders for each SCV measure made and the number of low-value orders for each SCV measure made. Carilion (and the other 7 participating health systems) are asked to use this information to generate quality improvement initiatives. We have designed a quality improvement initiative focused on family and community medicine clinicians and the two back pain measures.

First, we will use the most recent data provided by the SCV project (2020 and Q1-Q2 of 2021) to rank FCM practices and clinicians by utilization of low-value back pain services, their waste index, and impact score. We will identify from this ranking the top 5 to 10 performing practices and the bottom 5 to 10 performing practices. If there are any outlier clinicians who are bottom performing (ie: provide the most low-value services or have the highest impact score) but who do not fall among the bottom performing practices, we will consider including their practice among the bottom 5 to 10.

We will survey clinicians in top and bottom performing practices to learn more about their knowledge, perceptions, and practice workflow related to the two back pain measures. They will also be asked about their trust in data measures. No identifying information will be collected from clinicians in the survey.

From what we learn from survey data, we will design up to four brief education points to be communicated during regular practice quality improvement meetings with population health managers.

Prior to the delivery of quality improvement education about back pain measures, we will obtain an EMR report for the top and bottom performing practices showing utilization rate of both back pain measures. We will also conduct a chart review (Epic) to identify indication for provision of the back pain services that could not be detected in claims data or Epic data. This addresses a common concern of clinicians - that clinical nuance is not being detected and low value care is being over-assigned. The Epic reports and chart reviews will continue monthly for the first 3 months and then at months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

Current primary care clinician in a top or bottom performing practice

Exclusion Criteria:

<90 days of tenure in current position

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinicians (physicians, PAs, NPs)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge, perceptions, decision-making related to back pain imaging | June-August 2022
  Survey responses
Rate of low-value back pain imaging | June-August 2022
  Derived from APC data, via Milliman Health Waste Calculator
Rate of low-value back pain imaging | August 2022-December 2023
  Derived from EMR measures (live)
Clinical documentation comparison | August 2022-December 2023
  Comparison of EMR chart review reason for ordering imaging vs. EMR-derived measure

CONTACTS AND LOCATIONS:
Locations (1):
- Carilion Clinic Dept of Family and Community Medicine, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.

REFERENCES:
- See also: Related Info — https://www.vahealthinnovation.org/scv/